CLINICAL TRIAL: NCT02362425
Title: Antioxidant Therapy in RYR1-Related Congenital Myopathy
Acronym: RYR1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 150072; 15-NR-0072
Record Dates: First submitted 2015-02-12; First posted 2015-02-13 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-10-05

CONDITIONS: Neuromuscular Disease
Keywords: Neuromuscular Disease; Clinical Trial; Ryanodine Receptor Type 1; Myopathy
MeSH Terms: conditions — Neuromuscular Diseases; Muscular Diseases | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (3):
- RYR1-RM Patients Administered N-acetylcysteine (Active Comparator): N-acetylcysteine
  Interventions: Drug: N-acetylcysteine
- RYR1-RM Patients Administered Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Healthy Volunteers (No Intervention): Healthy volunteers who had physical exam, study biomarker, Near Infrared Spectroscopy (NIRS) testing and muscle ultrasound only, in one visit.

INTERVENTIONS:
Drug: N-acetylcysteine
  Arms: RYR1-RM Patients Administered N-acetylcysteine
Drug: Placebo
  Arms: RYR1-RM Patients Administered Placebo

SUMMARY:
Background:

- Ryanodine receptor type 1-related myopathies (RYR1-RM) are the most common non-dystrophic muscle diseases that people are born with in the U.S. They affect development, muscles, and walking. Researchers want to test a new drug to help people with these diseases.

Objectives:

- To see if the drug N-acetylcysteine decreases muscle damage in people with RYR1-RM. To see if it improves their exercise tolerance.

Eligibility:

- People age 7 and older with a confirmed genetic diagnosis of RYR1 or a clinical diagnosis of RYR1 and a family member with a confirmed genetic diagnosis.

Design:

* Participants will be screened with a checklist of criteria. Adult participants may have a muscle biopsy. A needle will remove a tiny piece of muscle in the lower leg.
* Study visits will take several days.
* Visit 1:
* Medical history
* Physical exam
* Blood, urine, and saliva tests
* Questions about symptoms and quality of life
* Heart, lung, and walking tests
* Muscle Oxygenation Capacity Test. A blood pressure cuff around the thigh will be tightened for up to 10 minutes.
* Biodex testing, stretching the leg against resistance
* Muscle ultrasounds. A probe will be moved over the skin.
* Participants may be photographed or videotaped during procedures.
* They may have a muscle biopsy.
* Six months later, visit 2 will repeat visit 1. Participants will start taking the study drug dissolved in water or placebo three times a day for 6 months.
* Participants will stay at NIH for 2 days after starting the study drug.
* Participants will be contacted by phone during the study to monitor side effects
* Six months after starting the study drug, study visit 3 will repeat some or all of visit 1.

DETAILED DESCRIPTION:
Although genetic disorders of muscle that present at birth are rare, RYR1-related myopathies comprise the most common non-dystrophic congenital myopathy in the United States, with a prevalence of approximately 1/90,000 people (Amburgey et al, 2011). Causative mutations in the ryanodine receptor gene of skeletal muscle, RYR1, have been found in several myopathy subtypes, including central core disease and centronuclear myopathy. These mutations result in defective excitation-contraction coupling and increased mitochondrial oxidative stress. Most patients present in childhood with delayed motor milestones, extremity muscle weakness, impaired ambulation, joint contractures, progressive scoliosis, and in some cases eye movement paralysis, respiratory failure, or susceptibility to malignant hyperthermia, an allelic condition. Despite these important morbidities and the risk of early mortality, no treatments exist to date.

RYR1 encodes a homotetrameric transmembrane ion channel, RyR1, which resides on the terminal sarcoplasmic reticulum in close proximity to the T-tubule. By releasing calcium from the sarcoplasmic reticulum into the cytosol in response to muscle fiber stimulation by the motor neuron at the neuromuscular junction, it mediates excitation-contraction coupling and functions as a regulator of cellular calcium concentrations and redox homeostasis. Dowling et al. (2012) recently elucidated the latter mechanism in zebrafish and patient myotubes, showing that RYR1 mutations result in increased oxidative stress and that this is rescued in both models by treatment with N-acetylcysteine (NAC), a known anti-oxidant. NAC functions as a precursor of glutathione, an endogenous antioxidant that becomes deficient during oxidative stress. This was substantiated by a cystic fibrosis clinical trial in which low glutathione levels in neutrophils undergoing oxidative stress significantly increased with NAC administration.

Dowling et al. (2012) found significant changes post NAC treatment including increased travel distance (endurance) in zebrafish and complete protection from cell death induced by experimentally increasing oxidative stress in myotubes. Thus NAC was a successful treatment in both ex vivo and in vivo model systems. Based on these results, we plan to perform a randomized, double-blinded, placebo controlled clinical trial of NAC in a subgroup of RYR1-related myopathy patients as the first pathophysiologically based treatment for this devastating disorder.

The objectives of the study are to determine if NAC reduces oxidative stress, fatigability, and fatigue in a study population of patients with RYR1-RM. The study population includes both males and females 7 years of age and older. The study design has two phases. The first 6-month phase will be used to validate the selected outcome measures in RYR1 congenital myopathy. The second 6-month phase is a randomized, double-blinded, placebo controlled drug intervention trial. The primary outcome measures are blood glutathione for oxidative stress and six minute walk test for fatigability. Healthy volunteers will be evaluated to determine normal values of biomarkers, muscle ultrasound, and near infrared spectroscopy in this rare disease, in order to develop a comparison between healthy and RYR1-RM individuals.

ELIGIBILITY:
* EXCLUSION CRITERIA - PATIENTS:
* Adults who cannot provide their own consent and pediatric participants who do not have a parent able to provide consent.
* Patients with a history of liver disease (Liver Function Tests will be collected at baseline and

at each study visit as a precautionary measure). Liver disease is defined as moderate to severe hepatic impairment based on the following:

* Alanine Aminotransferase (ALT) greater than or equal to 8x upper limit of normal (ULN) with total bilirubin 2x ULN (plus >35% direct bilirubin) and/or International normalized ratio (INR) >1.5 or
* Gamma-glutamyl transferase (GGT) > 2-3x ULN with bilirubin 2x ULN (plus >35% direct bilirubin) and/or INR

  * Patients with a history of peptic ulcers, gag reflex depression, and esophageal varices. Patients with gastrostomy tubes may be considered for participation, in the case of gag reflex depression or other swallowing or feeding difficulties.
  * Patients who have a severe pulmonary dysfunction (FEV1< 40% predicted) or evidence of pulmonary exacerbation. Pulmonary exacerbations refer to an acute worsening of respiratory symptoms that result from a decline in lung function. Participants may present with increased coughing, increased dyspnea, increased haemoptysis, increased fatigue, decreased pulmonary function by a min of 10%, or a change in sputum color.
  * Pregnant and breastfeeding women.
  * Consumption of antioxidants [including NAC, GSH, melatonin, Immunocal (Immunotac

Research, Vandreuil-Dorion, QC, Canada), Nacystelyn (Galephar, Brussels)] in the 4 weeks before recruitment.

-Daily use of acetaminophen (including Percocet, Vicodin, Oxycodone, Excedrin, and other

acetaminophen-containing drugs), nitroglycerine, or carbamazepine during the past 7 days.

* Current use of Angiotensin-converting enzyme (ACE) inhibitors or Angiotensin Receptor Blockers (ARBs).
* Patients who have ever used Beta2-adrenergic agonist tablets, for the purpose of increasing muscle mass (such as albuterol tablets).
* For the muscle biopsy procedure only (second and third visits, if applicable): Patients who have taken Aspirin, Ibuprofen, Advil, Motrin, or Aleve within the 3 days prior to the muscle biopsy procedure, and/or patients who have taken Plavix, fresh garlic, gingko, or ginseng 5 days prior to the muscle biopsy.
* Participation in trials for other therapeutic investigational drugs simultaneously or 4 weeks before recruitment.
* Other clinically significant medical disease that, in the judgment of the investigators, would expose the patient to undue risk of harm or prevent the patient from completing the study. Examples include anemia (defined as Hgb < 8 gm/dl), an inability to walk safely without assistance for at least 6 minutes, and/or an inability to consume at least 6 ounces of fluid, 3 times a day, either orally or via G-tube. Patients with comorbidities (i.e. cancer, epilepsy) will be carefully assessed to determine if their comorbidity could lead to confounding or safety issues, should their participation continue.

EXCLUSION CRITERIA - HEALTHY VOLUNTEERS:

* Diagnosis of RYR1-related myopathy or other neurological disorder (by neurological exam, genetic testing, or muscle biopsy
* Complaints of fatigue or weakness
* Consumption of antioxidants [including NAC, GSH, melatonin, Immunocal (Immunotac
* Research, Vandreuil-Dorion, QC, Canada), Nacystelyn (Galephar, Brussels)] in the 4 weeks before recruitment.
* Use of Beta2-adrenergic agonists.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-02-12; Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne J Wingate, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Chin LMK, Todd JJ, Chrismer IC, Witherspoon JW, Jain M, Waite M, Meilleur KG, Drinkard B, Lawal TA. Exercise capacity in RYR1-related myopathies. Orphanet J Rare Dis. 2025 Sep 24;20(1):485. doi: 10.1186/s13023-025-04013-7. PMID 40993798
- [Derived] Greer LK, Meilleur KG, Harvey BK, Wires ES. Identification of ER/SR resident proteins as biomarkers for ER/SR calcium depletion in skeletal muscle cells. Orphanet J Rare Dis. 2022 Jun 13;17(1):225. doi: 10.1186/s13023-022-02368-9. PMID 35698232
- [Derived] Todd JJ, Lawal TA, Witherspoon JW, Chrismer IC, Razaqyar MS, Punjabi M, Elliott JS, Tounkara F, Kuo A, Shelton MO, Allen C, Cosgrove MM, Linton M, Michael D, Jain MS, Waite M, Drinkard B, Wakim PG, Dowling JJ, Bonnemann CG, Emile-Backer M, Meilleur KG. Randomized controlled trial of N-acetylcysteine therapy for RYR1-related myopathies. Neurology. 2020 Mar 31;94(13):e1434-e1444. doi: 10.1212/WNL.0000000000008872. Epub 2020 Jan 15. PMID 31941795
- [Derived] Witherspoon JW, Vasavada RP, Waite MR, Shelton M, Chrismer IC, Wakim PG, Jain MS, Bonnemann CG, Meilleur KG. 6-minute walk test as a measure of disease progression and fatigability in a cohort of individuals with RYR1-related myopathies. Orphanet J Rare Dis. 2018 Jul 3;13(1):105. doi: 10.1186/s13023-018-0848-9. PMID 29970108
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-NR-0072.html

RESULTS

PARTICIPANT FLOW:
Groups:
- RYR1-RM Volunteers: Subjects with RYR1-RM entered into the Natural History Phase of the study.
- Healthy Volunteers: Healthy volunteers entered into the study for a one-visit assessment; no treatment given.
- RYR1-RM Volunteers: N-acetylcysteine (NAC): RYR1-RM subjects who were eventually randomized to NAC 900 mg tablets
- RYR1-RM Volunteers: Placebo: RYR1-RM subjects who were eventually randomized to Placebo 900 mg tablets without active NAC
Period: Phase 1 (up to 6 Months)
Arm/Group | RYR1-RM Volunteers | Healthy Volunteers | RYR1-RM Volunteers: N-acetylcysteine (NAC) | RYR1-RM Volunteers: Placebo
Started | 53 | 10 | 0 | 0
Completed | 37 | 10 | 0 | 0
Not Completed | 16 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Medicinal contraindication | 1 | 0 | 0 | 0
Not completed — Screening failure | 1 | 0 | 0 | 0
Not completed — Confirmatory genetic testing negative | 3 | 0 | 0 | 0
Not completed — Study closure | 9 | 0 | 0 | 0
Period: Phase 2 (up to 6 Months, Randomized)
Arm/Group | RYR1-RM Volunteers | Healthy Volunteers | RYR1-RM Volunteers: N-acetylcysteine (NAC) | RYR1-RM Volunteers: Placebo
Started | 0 | 0 | 16 | 17
Completed | 0 | 0 | 15 | 14
Not Completed | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Discontinued study drug due to procedure | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population contains the healthy volunteer participants, who only had one visit to determine normal values of biomarkers, muscle ultrasound, and near infrared spectroscopy in this rare disease, in order to develop a comparison between healthy and RYR1-RM individuals.
Groups:
- RYR1-RM Volunteers: All participants with RYR1-RM enrolled into the natural history period of the trial.
- Healthy Volunteers: Healthy volunteers were evaluated to determine normal values of biomarkers, muscle ultrasound, and near infrared spectroscopy in this rare disease, in order to develop a comparison between healthy and RYR1-RM individuals.
- RYR1-RM Volunteers: N-acetylcysteine (NAC): N-acetylcysteine (NAC) 900 mg tablets; week 1 up to 1800 mg/day; Week 2- through end of study based on participant weight: < 50 kg subjects up to 2700 mg/day, >50 kg subjects 2700 mg/day
- RYR1-RM Volunteers :Placebo: Placebo 900 mg tablets identical but did not contain NAC
- Total: Total of all reporting groups
Arm/Group | RYR1-RM Volunteers | Healthy Volunteers | RYR1-RM Volunteers: N-acetylcysteine (NAC) | RYR1-RM Volunteers :Placebo | Total
Number analyzed (Participants) | 53 | 10 | 16 | 17 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline measures are provided for the 53 RYR1-RM participants and the 10 healthy volunteers in the natural history phase, and for the 33 subjects who continued on into the randomized phase.
  years
    Phase 1: Natural History Period: number analyzed (Participants) | 53 | 10 | 0 | 0 | 63
    Phase 1: Natural History Period | 29.2 (17.5) | 44.8 (13.2) |  |  | 31.7 (17.9)
    Phase 2: Randomized Period: number analyzed (Participants) | 0 | 0 | 16 | 17 | 33
    Phase 2: Randomized Period |  |  | 28.1 (17.4) | 26.7 (18.5) | 27.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline measures are provided for the 53 RYR1-RM participants and the 10 healthy volunteers in the natural history phase, and for the 33 subjects who continued on into the randomized phase.
  Participants
    Phase 1: Natural History Period: number analyzed (Participants) | 53 | 10 | 0 | 0 | 63
    Phase 1: Natural History Period: Female | 29 | 7 |  |  | 36
    Phase 1: Natural History Period: Male | 24 | 3 |  |  | 27
    Phase 2: Randomized Period: number analyzed (Participants) | 0 | 0 | 16 | 17 | 33
    Phase 2: Randomized Period: Female |  |  | 9 | 10 | 19
    Phase 2: Randomized Period: Male |  |  | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline measures are provided for the 53 RYR1-RM participants and the 10 healthy volunteers in the natural history phase, and for the 33 subjects who continued on into the randomized phase.
  Participants
    Phase 1: Natural History Period: number analyzed (Participants) | 53 | 10 | 0 | 0 | 63
    Phase 1: Natural History Period: American Indian or Alaska Native | 0 | 0 |  |  | 0
    Phase 1: Natural History Period: Asian | 0 | 0 |  |  | 0
    Phase 1: Natural History Period: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Phase 1: Natural History Period: Black or African American | 6 | 2 |  |  | 8
    Phase 1: Natural History Period: White | 47 | 8 |  |  | 55
    Phase 1: Natural History Period: More than one race | 0 | 0 |  |  | 0
    Phase 1: Natural History Period: Unknown or Not Reported | 0 | 0 |  |  | 0
    Phase 2: Randomized Period: number analyzed (Participants) | 0 | 0 | 16 | 17 | 33
    Phase 2: Randomized Period: American Indian or Alaska Native |  |  | 0 | 0 | 0
    Phase 2: Randomized Period: Asian |  |  | 0 | 0 | 0
    Phase 2: Randomized Period: Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0
    Phase 2: Randomized Period: Black or African American |  |  | 1 | 0 | 1
    Phase 2: Randomized Period: White |  |  | 15 | 17 | 32
    Phase 2: Randomized Period: More than one race |  |  | 0 | 0 | 0
    Phase 2: Randomized Period: Unknown or Not Reported |  |  | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: This measure of Region of Enrollment is presented for subjects enrolled in the Natural History phase of the study as well as the Healthy Volunteers.
  Participants
    United States: number analyzed (Participants) | 53 | 10 | 0 | 0 | 63
    United States | 53 | 10 | 0 | 0 | 63
Region of Enrollment [Number; unit: participants] — Population: This measure of Region of Enrollment is presented for the subjects in the randomized period of the study, ie, randomized population.
  participants
    United States: number analyzed (Participants) | 0 | 0 | 16 | 17 | 33
    United States |  |  | 16 | 17 | 33
Body Mass Index BMI(kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline measures are provided for the 53 RYR1-RM participants and the 10 healthy volunteers in the natural history phase, and for the 33 subjects who continued on into the randomized phase.
  kg/m^2
    Phase 1: Natural History Period: number analyzed (Participants) | 53 | 10 | 0 | 0 | 63
    Phase 1: Natural History Period | 22.1 (8.7) | 32.1 (6.1) |  |  | 24.4 (8.7)
    Phase 2: Randomized Period: number analyzed (Participants) | 0 | 0 | 16 | 17 | 33
    Phase 2: Randomized Period |  |  | 22.8 (8.2) | 21.5 (6.5) | 21.9 (7.5)
Mode of Inheritance, dominant/de novo [Count of Participants; unit: Participants] — Mode of Inheritance is not applicable to healthy volunteer participants and therefore was not collected. Population: Mode of Inheritance is not applicable to healthy volunteer participants and therefore was not collected. Baseline measures are provided for each of the other two parts of the study: natural history and randomized. Of the 53 participants in the natural history period, 33 continued on into the randomized phase.
  Participants
    Phase 1: Natural History Period: number analyzed (Participants) | 53 | 0 | 0 | 0 | 53
    Phase 1: Natural History Period | 40 |  |  |  | 40
    Phase 2: Randomized Period: number analyzed (Participants) | 0 | 0 | 16 | 17 | 33
    Phase 2: Randomized Period |  |  | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Urine 15-F2t Isoprostane Concentration
Description: Urine will be assayed for 15-isoprostane-F2, which is formed when arachidonic acid reacts with reactive oxygen species(ROS). A validated gas chromatography(GC)-mass spectrometer (MS) method will be used to quantify 15-isoprostane-F2
Time Frame: 12 months
Population: Outcome measures are reported for participants who were randomized and continued into the randomized, double-blind period of the trial. Missing data was not imputed. This measure was not collected for Healthy Volunteers post-baseline (months 6 and 12), thus they are not included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mg Cr
Groups:
- N-acetylcysteine (NAC): N-acetylcysteine (NAC) 900 mg tablets; week 1 up to 1800 mg/day; Week 2- through end of study based on subject weight: < 50 kg subjects up to 2700 mg/day, >50 kg subjects 2700 mg/day
- Placebo: Placebo 900 mg tablets identical but did not contain NAC
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
ng/mg Cr | 2.7 [1.7 to 3.7] | 2.6 [1.5 to 3.6]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Null Hypothesis: In RYR1-RM myopathy patients, there will be no statistically significant difference in corrected 15-F2t-isoprostane concentration and/or corrected 15=f2t-Isop:PGR2alpha ratio between NAC and placebo groups at month 12, after controlling for established a priori confounders; Test type: Superiority — An a priori power calculation, with power at 80% and a two-sided α of 0·05, determined that n=76 participants (n=38 per group) would be required to detect a statistically significant post-intervention difference in plasma glutathione (GSH) concentration between NAC and placebo groups. After the primary endpoint was changed, re-evaluation of the sample size determined that a larger sample (total n=182) would be required. As per protocol, the study was completed at this time; p = 0.88, Regression, Linear; Model comparing 12 m corrected 15-F2t-isoprostane conc. controlling for pre-intervention value. Investigated covariates: smoking and drinking status; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.4 to 1.6]

2. Primary Outcome: Six Minute Walk Test (6MWT)
Description: Meters walked in 6 minutes will be recorded; distances in meters will be recorded at each minute interval; speed will be calculated.
Time Frame: 12 months
Population: Outcome measures are reported for participants who were randomized and continued into the randomized, double-blind period of the trial. Missing data was not imputed. This measure was not collected for Healthy Volunteers, thus they are not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
meters | 495.8 [475.8 to 515.9] | 471.9 [451.1 to 492.7]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; In RYR1-RM myopathy patients, there will be no statistically significant difference in 6MWT (six minute walk test) total distance between NAC and placebo groups at month 12, after controlling for established a priori confounders; Test type: Superiority; p = .11, Regression, Linear — Model controlled for six-month(pre-intervention) distance and treatment group. Investigated covariates: height; Mean Difference (Final Values) = 23.9, 95% CI 2-sided [-5.5 to 53.4]

3. Secondary Outcome: DCF-fluorescence Intensity (AU)
Description: Dichlorodihydrofluorescein (DCFH) will be used on participate muscle biopsies to analyze intracellular oxidant activity [H2DCFDA (H2-DCF, DCF)].
Time Frame: 12 months
Population: This analysis was performed only on participants in the randomized population who volunteered to have the muscle biopsy performed. This measure was not collected for Healthy Volunteers, thus they are not included in this analysis.
Measure: Mean (95% Confidence Interval); unit: AU
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 6 | 4
AU | 1.9 [0.7 to 3.1] | 3.4 [1.7 to 5.1]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.14, Regression, Linear; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-3.6 to 0.7]

4. Secondary Outcome: Time to Ascend Steps (Seconds)
Description: Participants completed the following timed function tests: supine to stand, ascend four steps, descend four steps, and walk/run 10 meters. For time taken to ascend four steps, the subject was asked to ascend four steps whilst being timed.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
seconds | 3.2 [2.9 to 3.5] | 3.3 [3.0 to 3.6]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.62, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.5 to 0.3]

5. Secondary Outcome: Descend Steps
Description: Participants completed the following timed function tests: supine to stand, ascend four steps, descend four steps, and walk/run 10 meters. For time taken to descend four steps, the subject was asked to descend four steps whilst being timed.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
seconds | 1.9 [1.5 to 2.3] | 2.4 [2.1 to 2.8]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.0]

6. Secondary Outcome: Walk/Run 10 Meters
Description: Participants completed the following timed function tests: supine to stand, ascend four steps, descend four steps, and walk/run 10 meters. For walk/run 10 meters, participants were timed as they walked/ran a marked 10-meter course as quickly as possible.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
seconds | 5.2 [4.3 to 6.1] | 5.9 [5.0 to 6.9]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.25, t-test, 2 sided; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-2.1 to 0.6]

7. Secondary Outcome: Supine to Stand
Description: Participants completed the following timed function tests: supine to stand, ascend four steps, descend four steps, and walk/run 10 meters. For time taken to transition from supine to standing, participants were asked to lay supine and then the time taken to move from supine to standing was recorded.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
seconds | 7.4 [6.6 to 8.1] | 8.4 [7.7 to 9.2]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-2.1 to 0.0]

8. Secondary Outcome: Motor Function Measure-32 (MFM-32) Domain 1 (D1)
Description: Motor Function Measure, MFM-32 is a well-established scale of motor function in congenital muscle disease. The D1 domains measure standard and transfers, and consist of 13 items. Generic Values for each domain are: 0 = cannot perform the task, 1 = initiated the task, 2 - performs the movement incompletely, or completely but imperfectly, 3 = performs the task fully and 'normally'. Total score is the sum of all the domains for D1 divided by the maximum score possible and multiplied by 100. Min=0, Max = 100. Lower numbers on the scale represent a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
% of maximum score | 74.9 [72.1 to 77.6] | 71.5 [68.6 to 74.3]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-0.6 to 7.3]

9. Secondary Outcome: Motor Function Measure-32 (MFM-32) Domain 2 (D2)
Description: Motor Function Measure, MFM-32 is a well-established scale of motor function in congenital muscle disease. The D2 domains measure axial and proximal motor function and consists of 12 items. Generic Values for each domain are: 0 = cannot perform the task, 1 = initiated the task, 2 - performs the movement incompletely, or completely but imperfectly, 3 = performs the task fully and 'normally'. The total score is the sum of all the MFM-32 domains for D2, divided by maximum score possible and multiplied by 100. Min = 0, Max = 100. Lower numbers on the scale represent a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
% of maximum score | 97.0 [95.9 to 98.1] | 96.7 [95.5 to 97.9]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.69, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.3 to 2.0]

10. Secondary Outcome: Motor Function Measure-32 (MFM-32) Domain 3 (D3)
Description: Motor Function Measure, MFM-32 is a well-established scale of motor function in congenital muscle disease. The D3 domains measure distal motor function and consist of 7 items. Generic Values for each domain are: 0 = cannot perform the task, 1 = initiated the task, 2 - performs the movement incompletely, or completely but imperfectly, 3 = performs the task fully and 'normally'. The total score is the sum of all the MFM-32 domains for D3, divided by maximum score possible and multiplied by 100. Min = 0, Max = 100. Lower numbers on the scale represent a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
% of maximum score | 95.5 [93.9 to 97.1] | 96.7 [95.0 to 98.3]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.31, t-test, 2 sided; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.5 to 1.1]

11. Secondary Outcome: Motor Function Measure-32 (MFM-32) Total Score
Description: Motor Function Measure, MFM-32 is a well-established scale of motor function in congenital muscle disease. Generic Values for each domain are: 0 = cannot perform the task, 1 = initiated the task, 2 - performs the movement incompletely, or completely but imperfectly, 3 = performs the task fully and 'normally'. The total score is the sum of all the MFM-32 domains, divided by maximum score possible (96) and multiplied by 100. Min = 0, Max = 100. Lower numbers on the scale represent a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
% of maximum score | 84.1 [82.8 to 85.4] | 83.0 [81.7 to 84.3]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.22, t-test, 2 sided; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.8 to 3.0]

12. Secondary Outcome: Hand Grip Strength
Description: Grip and pinch strength were determined using Myotools dynamometry. The myogrip hand held dynamometer was used to assess grip strength. Higher scores represent better outcomes.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
kg | 17.8 [16.1 to 19.5] | 17.9 [16.1 to 19.7]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.93, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-2.6 to 2.4]

13. Secondary Outcome: Hand Pinch Strength
Description: Grip and pinch strength were determined using Myotools dynamometry. The myopinch pinch gauge was used to measure finger strength. Higher scores represent better outcomes.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 15 | 14
kg | 4.7 [4.0 to 5.5] | 4.9 [4.2 to 5.7]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.66, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.3 to 0.8]

14. Secondary Outcome: Peak Torque Flexion
Description: Lower-body isometric strength testing was used to determine peak torque during flexion and extension. Participant's blood pressure was assessed, to rule-out hypertension (>140/90), prior to starting the test. Participants were then asked to push against a stationary arm and remained at the same joint angle for the duration of each test. Two short trials were completed to establish maximal force for each participant. This was followed by a long trial of flexion and extension to capture rate of fatigue to 50% after reaching their pre-determined maximal force. In the interest of safety, participants with hypertension and/or a history of knee injury did not perform the test.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
nM | 24.7 [23.0 to 26.3] | 22.6 [20.8 to 24.3]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-0.4 to 4.6]

15. Secondary Outcome: Peak Torque Extension
Description: as for outcome 14
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nM
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
nM | 24.7 [23.0 to 26.3] | 38.8 [35.3 to 42.2]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-0.7 to 9.0]

16. Secondary Outcome: Adult Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue
Description: Participants were asked to complete the PROMIS (patient-reported outcomes measurement information system) through the NIH online, self-administered Clinical Trials Survey System. PROMIS scores are normed to 100 meaning that the raw score is converted to a scale where 50 is the mean and the standard deviation is 10. Scores less than 50 indicate less fatigue compared to the average and scores over 50 indicate more fatigue than the average. Lower scores represent better outcomes.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 9 | 7
t score | 49.5 [43.9 to 55.1] | 55.0 [49.5 to 60.6]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.15, t-test, 2 sided; Mean Difference (Final Values) = -5.5, 95% CI 2-sided [-13.4 to 2.4]

17. Secondary Outcome: Adult Quality of Life in Neurological Disorders (NeuroQoL) Fatigue
Description: Participants were asked to complete the NeuroQoL questionnaire through the NIH online, self-administered Clinical Trials Survey System. The NeuroQoL scores were normed to 100, meaning that the raw score is converted to a scale where 50 is the mean and the standard deviation is 10. Scores less than 50 indicate less fatigue compared to the average and scores over 50 indicate more fatigue than the average. Lower scores represent better outcomes.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 9 | 7
t score | 45.1 [40.0 to 50.3] | 51.5 [46.3 to 56.6]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = -6.4, 95% CI 2-sided [-13.7 to 1.0]

18. Secondary Outcome: Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue
Description: Participants were asked to complete the PROMIS questionnaire through the NIH online, self-administered Clinical Trials Survey System. PROMIS scores were normed to 100 meaning that the raw scores were converted to a scale where 50 is the mean and the standard deviation is 10. Scores less than 50 indicate less fatigue compared to the average and scores over 50 indicate more fatigue than the average. Lower scores represent better outcomes.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 2 | 5
t score | 34.8 [18.5 to 88.2] | 51.1 [30.9 to 71.3]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.39, t-test, 2 sided; Mean Difference (Final Values) = -16.27, 95% CI 2-sided [-80.1 to 47.5]

19. Secondary Outcome: Pediatric Quality of Life in Neurological Disorders (NeuroQoL) Fatigue
Description: Participants were asked to complete the NeuroQoL questionnaire through the NIH online, self-administered Clinical Trials Survey System. NeuroQoL scores were normed to 100 meaning that the raw score is converted to a scale where 50 is the mean and the standard deviation is 10. Scores less than 50 indicate less fatigue compared to the average and scores over 50 indicate more fatigue than the average. Lower scores represent better outcomes.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 2 | 5
t score | 43.1 [0.7 to 85.5] | 53.1 [40.4 to 65.9]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.57, t-test, 2 sided; Mean Difference (Final Values) = 10.0, 95% CI 2-sided [-59.5 to 39.5]

20. Secondary Outcome: Multidimensional Fatigue Inventory - 20 (MFI-20) General Fatigue Score
Description: Participants were asked to complete the MFI-20 questionnaire through the NIH online, self-administered Clinical Trials Survey System. The MFI consists of 5 subscales: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation. Values range from 4-20 for each scale. Higher scores represent increased fatigue/ worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
scores on a scale | 11.6 [9.7 to 13.5] | 13.7 [11.7 to 15.8]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.12, t-test, 2 sided; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-5.0 to 0.6]

21. Secondary Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Physical Fatigue Score
Description: as for outcome 20
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
scores on a scale | 11.5 [9.3 to 13.6] | 11.9 [9.7 to 14.2]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.76, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-3.6 to 2.7]

22. Secondary Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Reduced Activity Score
Description: as for outcome 20
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
scores on a scale | 9.2 [7.2 to 11.2] | 8.7 [6.6 to 10.8]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.5 to 3.5]

23. Secondary Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Reduced Motivation Score
Description: as for outcome 20
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
scores on a scale | 7.8 [6.2 to 9.4] | 7.4 [5.7 to 9.1]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.70, t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.8 to 2.7]

24. Secondary Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Mental Fatigue Score
Description: as for outcome 20
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 14 | 12
scores on a scale | 8.8 [6.7 to 10.9] | 8.6 [6.4 to 10.8]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.88, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-2.8 to 3.3]

25. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Score
Description: Participants were asked to complete the FACIT-f questionnaire through the NIH online, self-administered Clinical Trials Survey System. Minimum value = 0, maximum value = 160. Higher scores represent a better outcome/ better QOL.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 9 | 7
scores on a scale | 76.1 [67.7 to 84.5] | 73.6 [64.1 to 83.2]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.61, t-test, 2 sided; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-10.3 to 15.2]

26. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Trial Outcome Index
Description: Participants were asked to complete the FACIT-F questionnaire through the NIH online, self-administered Clinical Trials Survey System. The Trial Outcome Index (TOI) is the sum of the physical well-being, functional well-being and 'additional concerns' subscales. The minimum value = 0, and maximum value = 52. Scores under 30 is considered to be severe fatigue. Higher scores represent a better outcome/QOL.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 9 | 7
scores on a scale | 37.6 [32.3 to 42.8] | 37.0 [31.0 to 42.9]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.87, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-7.4 to 8.5]

27. Secondary Outcome: Pediatric Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Score
Description: Pediatric participants (< 18 years) were asked to complete the Peds-FACIT-F questionnaire through the NIH online, self-administered Clinical Trials Survey System.Minimum value = 0, maximum value = 52. Higher scores represent a better outcome/ better QOL.
Time Frame: 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 6 | 6
scores on a scale | 29.8 [12.0 to 47.6] | 42.3 [30.4 to 54.3]
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority; p = 0.28, t-test, 2 sided; Mean Difference (Final Values) = -12.5, 95% CI 2-sided [-38.9 to 13.9]

28. Secondary Outcome: Blood Glutathione Reduced (GSH):Oxidized (GSSG) Ratio
Description: GSH:GSSG ratio analyzed only at baseline to offer comparison of RYR1-RM affected individuals to the general population.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Healthy Volunteer: Healthy volunteers who participated in a one-visit assessment.
Arm/Group | RYR1-RM Volunteers | Healthy Volunteer
Number analyzed (Participants) | 38 | 10
ratio | 10.8 (7.2) | 0.54 (1.18)

29. Other Pre Specified Outcome: Urine 15-F2t Isoprostane Concentration Pre-Intervention
Description: as for outcome 1
Time Frame: 6 months
Population: Outcome measures are reported for participants who were randomized and continued into the randomized, double-blind period of the trial. Missing data was not imputed. This measure was not collected for Healthy Volunteers post baseline, thus they are not included in this analysis..
Measure: Mean (Standard Deviation); unit: ng/mg Cr
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 16
ng/mg Cr | 3.6 (2.2) | 3.1 (1.9)

30. Other Pre Specified Outcome: Six Minute Walk Test (6MWT) Pre-Intervention
Description: as for outcome 2
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
meters | 519.1 (119.0) | 453.8 (128.5)

31. Other Pre Specified Outcome: DCF-fluorescence Intensity (AU) Pre-Intervention
Description: as for outcome 3
Time Frame: 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: AU
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 7 | 5
AU | 1.7 (0.9) | 2.0 (1.6)

32. Other Pre Specified Outcome: Time to Ascend Steps (Seconds) Pre-Intervention
Description: as for outcome 4
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
seconds | 2.9 (1.5) | 3.4 (1.8)

33. Other Pre Specified Outcome: Descend Steps Pre-Intervention
Description: as for outcome 5
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
seconds | 2.2 (1.0) | 2.3 (1.0)

34. Other Pre Specified Outcome: Walk/Run 10 Meters Pre-Intervention
Description: as for outcome 6
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 15
seconds | 5.0 (2.2) | 4.6 (1.7)

35. Other Pre Specified Outcome: Supine to Stand Pre-Intervention
Description: as for outcome 7
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 15
seconds | 6.9 (5.5) | 6.7 (5.4)

36. Other Pre Specified Outcome: Motor Function Measure-32 (MFM-32) Domain 1 (D1) Pre-Intervention
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
% of maximum score | 75.8 (16.6) | 71.6 (21.2)

37. Other Pre Specified Outcome: Motor Function Measure-32 (MFM-32) Domain 2 (D2) Pre-Intervention
Description: as for outcome 9
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
% of maximum score | 96.0 (4.8) | 96.6 (7.3)

38. Other Pre Specified Outcome: Motor Function Measure-32 (MFM-32) Domain 3 (D3) Pre-Intervention
Description: as for outcome 10
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
% of maximum score | 96.7 (3.8) | 95.2 (5.3)

39. Other Pre Specified Outcome: Motor Function Measure-32 (MFM-32) Total Score Pre-Intervention
Description: as for outcome 11
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % of maximum score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
% of maximum score | 84.4 (7.6) | 82.7 (9.8)

40. Other Pre Specified Outcome: Hand Grip Strength Pre-Intervention
Description: as for outcome 12
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
kg | 20.5 (14.0) | 17.5 (11.0)

41. Other Pre Specified Outcome: Hand Pinch Strength Pre-Intervention
Description: as for outcome 13
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 17
kg | 6.5 (5.0) | 5.1 (2.3)

42. Other Pre Specified Outcome: Peak Torque Flexion Pre-Intervention
Description: as for outcome 14
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 14
nM | 31.9 (22.0) | 25.2 (21.3)

43. Other Pre Specified Outcome: Peak Torque Extension Pre-Intervention
Description: as for outcome 14
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 16 | 14
nM | 56.9 (42.9) | 41.6 (45.5)

44. Other Pre Specified Outcome: Adult Patient-Reported Outcomes Measurement Information System (PROMIS) - Fatigue Pre-Intervention
Description: as for outcome 16
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 7 | 10
t score | 59.2 (11.8) | 58.5 (11.3)

45. Other Pre Specified Outcome: Adult Quality of Life in Neurological Disorders (NeuroQoL) Fatigue Pre-Intervention
Description: as for outcome 17
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 7 | 10
t score | 53.25 (8.5) | 51.9 (7.4)

46. Other Pre Specified Outcome: Pediatric Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Pre-Intervention
Description: as for outcome 18
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 4 | 4
t score | 42.6 (8.4) | 57.3 (7.7)

47. Other Pre Specified Outcome: Pediatric Quality of Life in Neurological Disorders (NeuroQoL) Fatigue Pre-Intervention
Description: as for outcome 19
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: t score
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 4 | 5
t score | 45.9 (6.4) | 52.8 (2.8)

48. Other Pre Specified Outcome: Multidimensional Fatigue Inventory - 20 (MFI-20) General Fatigue Score Pre-Intervention
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 13 | 15
scores on a scale | 12.9 (4.2) | 14.3 (3.8)

49. Other Pre Specified Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Physical Fatigue Score Pre-Intervention
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 13 | 15
scores on a scale | 12.1 (5.6) | 13.0 (3.9)

50. Other Pre Specified Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Reduced Activity Score Pre-Intervention
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 13 | 15
scores on a scale | 9.5 (4.7) | 11.3 (3.2)

51. Other Pre Specified Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Reduced Motivation Score Pre-Intervention
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 13 | 15
scores on a scale | 7.9 (3.1) | 9.1 (3.5)

52. Other Pre Specified Outcome: Multidimensional Fatigue Inventory-20 (MFI-20) Mental Fatigue Score Pre-Intervention
Description: as for outcome 20
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 13 | 15
scores on a scale | 8.8 (4.8) | 9.7 (4.4)

53. Other Pre Specified Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Score Pre-Intervention
Description: as for outcome 25
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 9 | 10
scores on a scale | 69.2 (16.9) | 71.3 (20.9)

54. Other Pre Specified Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Trial Outcome Index Pre-Intervention
Description: as for outcome 26
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 9 | 10
scores on a scale | 33.8 (11.4) | 34.3 (10.3)

55. Other Pre Specified Outcome: Pediatric Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Total Score Pre-Intervention
Description: as for outcome 27
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 5 | 4
scores on a scale | 43.2 (7.7) | 37.0 (8.4)

56. Other Pre Specified Outcome: Urine 15-F2t Isoprostane Concentration at Baseline
Description: as for outcome 1
Time Frame: Baseline
Population: Healthy volunteers who participated in a one-visit assessment and RYR1-RM Volunteers measured at Baseline.
Measure: Mean (Standard Deviation); unit: ng/mg Cr
Arm/Group | RYR1-RM Volunteers | Healthy Volunteers
Number analyzed (Participants) | 49 | 10
ng/mg Cr | 3.17 (1.48) | 1.36 (0.48)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from start of study drug through the end of the study at 12 months. AEs were analyzed for the natural history period and the treatment period separately.
Description: (Institutional Review Board) IRB determination was used for the classification of adverse events
Groups:
- RYR1-RM Volunteers: N-acetylcysteine (NAC): N-acetylcysteine (NAC) 900 mg tablets for 6 months; week 1 up to 1800 mg/day; Week 2- through end of study based on subject weight: < 50 kg subjects up to 2700 mg/day, >50 kg subjects 2700 mg/day
- RYR1-RM Volunteers :Placebo: Placebo 900 mg tablets for 6 months; identical but did not contain NAC
- Healthy Volunteers: Healthy volunteers were evaluated at a one-visit assessment at baseline to determine normal values of biomarkers, muscle ultrasound, and near infrared spectroscopy in order to develop a comparison between healthy and RYR1-RM individuals
Arm/Group | RYR1-RM Volunteers | RYR1-RM Volunteers: N-acetylcysteine (NAC) | RYR1-RM Volunteers :Placebo | Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/16 | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/53 | 4/16 | 5/17 | 0/10
Other Adverse Events (participants affected / at risk) | 36/53 | 16/16 | 17/17 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RYR1-RM Volunteers (N=53) | RYR1-RM Volunteers: N-acetylcysteine (NAC) (N=16) | RYR1-RM Volunteers :Placebo (N=17) | Healthy Volunteers (N=10)
Intestinal Malrotation (Congenital, familial and genetic disorders) | 1 | 1 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | NA
Uterine Leiomyoma (Reproductive system and breast disorders) | 0 | 0 | 1 | NA
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | NA
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | NA
Hypotension (Vascular disorders) | 0 | 1 | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RYR1-RM Volunteers (N=53) | RYR1-RM Volunteers: N-acetylcysteine (NAC) (N=16) | RYR1-RM Volunteers :Placebo (N=17) | Healthy Volunteers (N=10)
Blurred Vision (Eye disorders) | 0 | 1 | 0 | 0
Barrett's Oesophagus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Stomach Virus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 3 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Faecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 4 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Influenza-like Illness (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 2 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Gamma-glutamyl Transferase Increased (Investigations) | 1 | 2 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 1
Prothombin Time Prolonged (Investigations) | 0 | 0 | 2 | 0
Red Cell Distribution Width Increased (Investigations) | 1 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 | 0 | 1 | 0
Blood Creatinine Phosphokinase Increased (Investigations) | 0 | 0 | 1 | 0
Blood Creatinine Decreased (Investigations) | 5 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Enchondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 3 | 0
Memory Impairment (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Left inguinal lymph node (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Malrotation of bowel (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0
Hematocrit increased (Investigations) | 2 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 1 | 0 | 0 | 0
Mean corpuscular volume increased (Investigations) | 2 | 0 | 0 | 0
mean corpuscular hemoglobin concentration decreased (Investigations) | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 3 | 0 | 0 | 2
Creatinine kinase increased (Investigations) | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 2 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1
Arthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone island benign tumor (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine fibroids (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Mean Platelet Volume (MVP) low (Investigations) | 0 | 0 | 0 | 1
Bilirubin high (Investigations) | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT02362425/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT02362425/SAP_001.pdf